CLINICAL TRIAL: NCT04714437
Title: Relationship Between the Frequency of Masticatory Side Switches and Aspects of Masticatory Function.
Brief Title: Masticatory Side Change and Masticatory Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Jordi Martinez-Gomis, Associate Professor DDS. PhD, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HOUB 36/2020
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Chewing Problem; Mastication Disorder
Keywords: Chewing side; Masticatory side switch; Mastication; Masticatory rhythm; Masticatory performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- F-R/L-A1/A3/A5 Sequence (Active Comparator): First, 5 freestyle masticatory assays (F). Second, 5 only-right (R) and 5 only-left (L) masticatory assays in the following order (R-L-L-R-R-L-L-R-R-L) Third, 15 masticatory assays changing the side once (A1), three times (A3) or 5 times (A5) in the following order (A1-A3-A5-A5-A3-A1-A1-A3-A5-A5-A3-A1-A1-A3-A5)
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: A1; Behavioral: A3; Behavioral: A5
- F-R/L-A1/A5/A3 Sequence (Active Comparator): First, 5 freestyle masticatory assays (F). Second, 5 only-right (R) and 5 only-left (L) masticatory assays in the following order (R-L-L-R-R-L-L-R-R-L) Third, 15 masticatory assays changing the side once (A1), three times (A3) or 5 times (A5) in the following order (A1-A5-A3-A3-A5-A1-A1-A5-A3-A3-A5-A1-A1-A5-A3)
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: A1; Behavioral: A3; Behavioral: A5
- F-R/L-A3/A1/A5 Sequence (Active Comparator): First, 5 freestyle masticatory assays (F). Second, 5 only-right (R) and 5 only-left (L) masticatory assays in the following order (R-L-L-R-R-L-L-R-R-L) Third, 15 masticatory assays changing the side once (A1), three times (A3) or 5 times (A5) in the following order (A3-A1-A5-A5-A1-A3-A3-A1-A5-A5-A1-A3-A3-A1-A5)
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: A1; Behavioral: A3; Behavioral: A5
- F-R/L-A3/A5/A1 Sequence (Active Comparator): First, 5 freestyle masticatory assays (F). Second, 5 only-right (R) and 5 only-left (L) masticatory assays in the following order (R-L-L-R-R-L-L-R-R-L) Third, 15 masticatory assays changing the side once (A1), three times (A3) or 5 times (A5) in the following order (A3-A5-A1-A1-A5-A3-A3-A5-A1-A1-A5-A3-A3-A5-A1)
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: A1; Behavioral: A3; Behavioral: A5
- F-R/L-A5/A1/A3 Sequence (Active Comparator): First, 5 freestyle masticatory assays (F). Second, 5 only-right (R) and 5 only-left (L) masticatory assays in the following order (R-L-L-R-R-L-L-R-R-L) Third, 15 masticatory assays changing the side once (A1), three times (A3) or 5 times (A5) in the following order (A5-A1-A3-A3-A1-A5-A5-A1-A3-A3-A1-A5-A5-A1-A3)
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: A1; Behavioral: A3; Behavioral: A5
- F-R/L-A5/A3/A1 Sequence (Active Comparator): First, 5 freestyle masticatory assays (F). Second, 5 only-right (R) and 5 only-left (L) masticatory assays in the following order (R-L-L-R-R-L-L-R-R-L) Third, 15 masticatory assays changing the side once (A1), three times (A3) or 5 times (A5) in the following order (A5-A3-A1-A1-A3-A5-A5-A3-A1-A1-A3-A5-A5-A3-A1)
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: A1; Behavioral: A3; Behavioral: A5

INTERVENTIONS:
Behavioral: F — The participant will be asked to chew the latex bag naturally.
Behavioral: R — The participant will be asked to chew the latex bag unilaterally on the right-side.
Behavioral: L — The participant will be asked to chew the latex bag unilaterally on the left-side.
Behavioral: A1 — The participant will be asked to chew the latex bag changing the side once.
Behavioral: A3 — The participant will be asked to chew the latex bag changing the side three times.
Behavioral: A5 — The participant will be asked to chew the latex bag changing the side five times.

SUMMARY:
The primary objective of this study is to establish the effect of the frequency of masticatory side switches on masticatory performance. We also want to know the effect of the frequency of masticatory side switches on the masticatory rhythm. Twenty-eight healthy volunteers will undertake masticatory tests, following a series of instructions given at the moment. These volunteers will take a re-test in two-weeks time. The sequence of these tests will be randomized in such a way that, each participant will initially perform an established sequence of "freestyle, only-right, and only-left" masticatory tests, and then will carry out one of the 6 possible combinations of "A1, A3, and A5". These tests will be recorded on video to assess, on slow playback, the change of the chewing side, and the masticatory rhythm.Masticatory performance will be determined by sieving the silicone particles.

DETAILED DESCRIPTION:
This crossover intervention study aims to assess the effect of the degree of alternance of the chewing side on various aspects of masticatory function, including masticatory performance and rhythm. Twenty-eight volunteers will take part, recruited for convenience, among friends and relatives of the teachers and students of the Degree of Dentistry of the Faculty of Medicine and Health Sciences of the University of Barcelona. These individuals will perform masticatory tests and, after a period of two weeks, will repeat them as a re-test. Each participant will perform 6 tests, each consisting of 5 assays, chewing a small latex bag containing a few silicone tablets (2 g) during 20 masticatory cycles. One test involves freestyle mastication in which the participant will be asked to chew the latex bag naturally. Two tests involve chewing the bag unilaterally (i.e., right-hand side in one and left-hand side in the other) and the order of their assays will be varied. For the last three tests, the participant will change the chewing side 1 (A1), 3 (A3), or 5 (A5) times respectively; the sequence of the assays will be randomized. The masticatory performance will be determined by the "median particle size" (MPS), and the masticatory rhythm will be assessed through the masticatory frequency as the ratio of masticatory cycle number to masticatory time. The control variables will include age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* Natural dentition (minimum 24 teeth).

Exclusion Criteria:

* Active orthodontics treatment.
* Intraoral pain.
* Temporomandibular joint pain.
* Masticatory muscle pain.
* Large dental restorations.
* Dental prosthesis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Masticatory performance | 1 hour 30 minutes
  The masticatory performance will be calculated for each test (free, only-right, only-left, and guided tests). The particles from the 5 assays (10g) will be allowed to dry for 24 h. They will then be passed through a series of 8 sieves of different sizes (sizes are: 0.25, 0.425, 0.85, 2, 2.8, 3.15, 4 and 5.6mm). To allow the particles to pass through the sieves, they will be stirred for 6 min. The weight of the remaining pieces of silicone in each sieve will be weighed and the "Median Particle Size" (MPS) will be calculated using the Rosin Rammler formula. The MPS or (X50) is the aperture in mm of a theoretic sieve through which 50% of the weight of the particles would pass, therefore, the smaller the value of MPS, the more masticatory performance the individual has.
Masticatory Frequency | 1 hour 30 minutes
  Masticatory frequency will be assessed as the ratio of masticatory cycle number to masticatory time (in cycles per minute).

SECONDARY OUTCOMES:
Side Switch Index | 1 hour 30 minutes
  The number of side switches during the 20 masticatory cycles for each assay will be determined using slow playback of the video recordings of the freestyle mastication test. In the case that this switch is a change of side from left to right or right to left, we will assign a value of "1". If this switch consists of a change from the right or left to central or vice versa, we will assign a value of "0.5". If there is no change of side, the value assigned to this chewing cycle will be "0". To determine the Side Switch Index, the number of side changes will be divided by the maximum number of changes possible during these 5 assays (95).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, University of Barcelona, L'Hospitalet de Llobregat, Catalonia, Spain

REFERENCES:
- [Background] Albert TE, Buschang PH, Throckmorton GS. Masticatory performance: a protocol for standardized production of an artificial test food. J Oral Rehabil. 2003 Jul;30(7):720-2. doi: 10.1046/j.1365-2842.2003.01155.x. PMID 12791158
- [Background] Buschang PH, Throckmorton GS, Travers KH, Johnson G. The effects of bolus size and chewing rate on masticatory performance with artificial test foods. J Oral Rehabil. 1997 Jul;24(7):522-6. doi: 10.1046/j.1365-2842.1997.00524.x. PMID 9250840
- [Background] Farias Gomes SG, Custodio W, Moura Jufer JS, Del Bel Cury AA, Rodrigues Garcia RC. Correlation of mastication and masticatory movements and effect of chewing side preference. Braz Dent J. 2010;21(4):351-5. doi: 10.1590/s0103-64402010000400011. PMID 20976387
- [Background] Flores-Orozco EI, Tiznado-Orozco GE, Osuna-Gonzalez OD, Amaro-Navarrete CL, Rovira-Lastra B, Martinez-Gomis J. Lack of relationship between masticatory performance and nutritional status in adults with natural dentition. Arch Oral Biol. 2016 Nov;71:117-121. doi: 10.1016/j.archoralbio.2016.07.008. Epub 2016 Jul 29. PMID 27494213
- [Background] Julien KC, Buschang PH, Throckmorton GS, Dechow PC. Normal masticatory performance in young adults and children. Arch Oral Biol. 1996 Jan;41(1):69-75. doi: 10.1016/0003-9969(95)00098-4. PMID 8833593
- [Background] Khoury-Ribas L, Ayuso-Montero R, Rovira-Lastra B, Peraire M, Martinez-Gomis J. Reliability of a new test food to assess masticatory function. Arch Oral Biol. 2018 Mar;87:1-6. doi: 10.1016/j.archoralbio.2017.12.006. Epub 2017 Dec 9. PMID 29241026
- [Background] Remijn L, Groen BE, Speyer R, van Limbeek J, Nijhuis-van der Sanden MW. Reproducibility of 3D kinematics and surface electromyography measurements of mastication. Physiol Behav. 2016 Mar 1;155:112-21. doi: 10.1016/j.physbeh.2015.11.018. Epub 2015 Nov 23. PMID 26617403
- [Background] Rovira-Lastra B, Flores-Orozco EI, Salsench J, Peraire M, Martinez-Gomis J. Is the side with the best masticatory performance selected for chewing? Arch Oral Biol. 2014 Dec;59(12):1316-20. doi: 10.1016/j.archoralbio.2014.08.005. Epub 2014 Aug 18. PMID 25173664
- [Background] Mioche L, Hiiemae KM, Palmer JB. A postero-anterior videofluorographic study of the intra-oral management of food in man. Arch Oral Biol. 2002 Apr;47(4):267-80. doi: 10.1016/s0003-9969(02)00007-9. PMID 11922870
- [Background] Khoury-Ribas L, Ignatova-Mishutina T, Rovira-Lastra B, Ayuso-Montero R, Martinez-Gomis J. Impact of Treatment with Unilateral Implant- Supported Fixed Partial Prosthesis on the Frequency of Masticatory Side Switches in Patients with Unilateral Posterior Missing Teeth. Eur J Prosthodont Restor Dent. 2022 Nov 30;30(4):245-251. doi: 10.1922/EJPRD_2336Khoury-Ribas07. PMID 35107226
- [Result] Ignatova-Mishutina T, Khoury-Ribas L, Flores-Orozco EI, Rovira-Lastra B, Martinez-Gomis J. Effect of side switch frequency on masticatory performance and rhythm in adults with natural dentition: A randomised crossover trial. J Oral Rehabil. 2022 Apr;49(4):373-380. doi: 10.1111/joor.13308. Epub 2022 Feb 12. PMID 35108409
- See also: Mizumori T, Arai K, Tsubakimoto T, Yatani H. Chewing side continuity and masticatory performance. Prosthodont Res Pract. 2006;5:10-4. — https://doi.org/10.2186/prp.5.10